CLINICAL TRIAL: NCT01365000
Title: A Phase I, Open-label, Randomized, Balanced, Single-dose, Two-Part Study to Assess the Relative Bioavailability of NKTR-118 in Three Formulations Under Fasted (3-Way Crossover) and Fed (2-Way Crossover) Conditions in Male and Non-fertile Female Subjects
Brief Title: Assessment of Relative Bioavailability of NKTR-118 in Three Formulations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D3820C00025
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Phase 1; Pharmacokinetics; NKTR-118; fasting or fed state; cross-over study; AUC(0-t); Cmax; tmax; QTcF Interval
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- NKTR118 Formulation 1 (Experimental): Fasted
  Interventions: Drug: NKTR118 Formulation 1
- NKTR118 Formulation 2 (Experimental): Fasted
  Interventions: Drug: NKTR118 Formulation 2
- NKTR118 Formulation 3 (Experimental): Fasted
  Interventions: Drug: NKTR118 Formulation 3
- NKTR118 Formulation 1a (Experimental): Fed
  Interventions: Drug: NKTR118 Formulation 1a
- NKTR118 Formulation 3a (Experimental): FED
  Interventions: Drug: NKTR118 Formulation 3a

INTERVENTIONS:
Drug: NKTR118 Formulation 1 — Oral dose, 25 mg
  Arms: NKTR118 Formulation 1
Drug: NKTR118 Formulation 2 — Oral dose, 25 mg
  Arms: NKTR118 Formulation 2
Drug: NKTR118 Formulation 3 — Oral dose, 25 mg
  Arms: NKTR118 Formulation 3
Drug: NKTR118 Formulation 1a — Oral dose, 25 mg
  Arms: NKTR118 Formulation 1a
Drug: NKTR118 Formulation 3a — Oral dose, 25 mg
  Arms: NKTR118 Formulation 3a

SUMMARY:
The is an assessment of Relative Bioavailability of NKTR-118 in Three Formulations in Healthy Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures
* Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating, and must be of non-childbearing potential, confirmed at screening by fulfilling one of the following criteria:
* Post-menopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and with follicle stimulating hormone (FSH) levels in the laboratory defined post-menopausal range
* Irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not tubal ligation
* Volunteers must have a body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg
* Volunteers must be able to understand and be willing to comply with study procedures, restrictions and requirements
* Healthy male and non-fertile female volunteers ages 18 to 55 years inclusive, with suitable veins for cannulation or repeated venipuncture

Exclusion Criteria:

* Any clinically significant disease or disorder (eg, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment) which, in the opinion of the Investigator, may either put the healthy volunteer at risk because of participation in the study, or influence the absorption, distribution, metabolism, and excretion of drugs
* Current smokers, those who have smoked or used nicotine products within the previous 3 months from the date of screening (Visit 1)
* Plasma donation within 1 month of screening or any blood donation/blood loss >500 mL during the 3 months prior to screening or intention to donate blood or blood products during the study or within 3 months after the completion of the study
* Positive screen for drugs of abuse, or cotinine (nicotine level above 400 ng/mL), at screening or admission and/or positive alcohol test at admission
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational product

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics after a dose of NKTR-118 25 mg by assessment of (Cmax) | day-1 to day 3
Pharmacokinetics after a dose of NKTR-118 25 mg by assessment of time to Cmax (tmax) | day-1 to day 3
Pharmacokinetics after a dose of NKTR-118 25 mg by assessment of half-life (t1/2λz) | day-1 to day 3
Pharmacokinetics after a dose of NKTR-118 25 mg by assessment of area under concentration-time curve (AUC(0-t)) | day-1 to day 3
Pharmacokinetics after a dose of NKTR-118 25 mg by assessment of area from time zero (pre-dose) extrapolated to infinity (AUC). | day-1 to day 3

SECONDARY OUTCOMES:
Safety and tolerability of NKTR-118 following administration of a single oral doses of NKTR-118 of 3 different formulations during fed and fasted conditions by assessing adverse events | Duration day -1 (Visit 2) to follow up (Visit 12)
Safety and tolerability of NKTR-118 following administration of a single oral doses of NKTR-118 of 3 different formulations during fed and fasted conditions by assessing Safety Laboratory values | Duration day -1 (Visit 2) to follow up (Visit 12)
Safety and tolerability of NKTR-118 following administration of a single oral doses of NKTR-118 of 3 different formulations during fed and fasted conditions by assessing 12-Lead Electrocardiograms | Duration day -1 (Visit 2) to follow up (Visit 12)
Safety and tolerability of NKTR-118 following administration of a single oral doses of NKTR-118 of 3 different formulations during fed and fasted conditions by assessing Columbia-Suicide Severity Rating Scale (C-SSRS) | Duration day -1 (Visit 2) to follow up (Visit 12)
Concentration of NKTR-118 in plasma samples after drug intake during Fed condition | Duration: Day 1 to day 4 at the 2 last inhouse stays

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, MD, Study Director — AstraZeneca; David Mathews, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- See also: D3820C00025 Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1399&filename=D3820C00025_Clinical_Study_Report_Synopsis.pdf